CLINICAL TRIAL: NCT05316181
Title: Randomized Phase III Trial of Cytoreductive Surgery (CRS) and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) for Platinum-Resistant Recurrent Ovarian Cancer: KOV-02R - Resistant Cancer of Ovary (RECOVER)
Brief Title: CRS & HIPEC for Platinum-Resistant Recurrent Ovarian Cancer (KOV-02R, RECOVER)
Acronym: KOV-HIPEC-02R
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Myong Cheol Lim, MD, PhD, Principal investigator, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC2021-0334
Record Dates: First submitted 2022-03-03; First posted 2022-04-07 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Epithelial Ovarian Cancer; Platinum Resistant; Recurrent Ovarian; HIPEC; Mitomycin; Cytoreductive Surgery
Keywords: Ovarian cancer; Hyperthermic intraperitoneal chemotherapy; HIPEC; Recurrent ovarian cancer; Cytoreductive surgery; Platinum-Resistant; Doxorubicin; Mitymycin
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled, open-label, multicenter phase III trial
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cytoreductive surgery and HIPEC (Experimental): Cytoreductive surgery + Hyperthermic Intraperitoneal Chemotherapy (HIPEC) followed by physician-choice chemotherapy until disease progression.
  Interventions: Procedure: HIPEC
- No HIPEC (No Intervention): Physician-choice chemotherapy from enrollment until disease progression.

INTERVENTIONS:
Procedure: HIPEC — HIPEC perfusion, doxorubicin 35mg/m2 & mitomycin 15 mg/m2, 41.5'C, 90 min.
  Arms: Cytoreductive surgery and HIPEC

SUMMARY:
Platinum-resistant recurrent epithelial ovarian cancer randomizing with or without cytoreductive surgery + hyperthermic intraperitoneal chemotherapy (HIPEC): KOV-02R, RECOVER

DETAILED DESCRIPTION:
The objective of this trial (KOV-HIPEC-02R) is to prove the survival benefit of HIPEC with doxorubicin and mitomycin (trial arm) compared to physician-choice chemotherapy (control arm) in patients with platinum-resistant recurrent epithelial ovarian cancer.

ELIGIBILITY:
* Inclusion Criteria:

  * Patients ≥18 years old,
  * Patients with Eastern Cooperative Oncology Group (ECOG) Performance status 0-2,
  * Patients diagnosed with histologically confirmed epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer,
  * Resistant to platinum-based chemotherapy (Platinum-refractory or resistant disease)
  * Resectable intraperitoneal disease based on previous clinical history and recent image finding,
  * A life expectancy > 3 months as clinically judged,
  * Women who are medically unable to conceive or who are of childbearing potential, agree to follow contraceptive guidelines during treatment,
  * Patient can also consent to the provision of clinical information for secondary use such as future biomedical research. However, in the future, subjects can participate in the main trial even if they do not intend to participate in sharing clinical information and,
  * Adequate organ function for cytoreductive surgery and HIPEC
* Exclusion criteria:

  * Non-epithelial ovarian carcinoma,
  * Borderline ovarian tumor,
  * Patients who are not appropriate for surgical and HIPEC procedures based on previous surgery or clinical findings, including severe intestinal adhesions, obstruction, or abdominal fistula,
  * Patients with myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with features suggestive of MDS/AML,
  * Patients which extra-abdominal disease is a major disease or is expected to cause of death,
  * Patients with active central nervous system metastasis and carcinoma meningitis or patients who have been previously treated for brain metastases must be in a stable state in radiology,
  * Patients with antibacterial, antifungal, or antiviral infections requiring systemic treatment (administration of parenteral antibiotics),
  * Active tuberculosis that is not controlled within 1 month of treatment,
  * Patient diagnosed with a psychiatric disorder or substance abuse disorder that would interfere with your ability to cooperate with the trial,
  * Patients who have not undergone hysterectomy and have a positive urine pregnancy test result within 14 days prior to clinical trial assignment, even if the urine pregnancy test result is negative at screening,
  * Pregnant or lactating women,
  * Patients with any contraindications to the use of doxorubicin or mitomycin (i.e., hypersensitivity to doxorubicin or mitomycin),
  * Patients with a history of allogeneic tissue/solid organ transplantation or bone marrow transplantation or a history of double umbilical cord transplantation or,
  * History or current evidence of any condition, therapy, or laboratory abnormality that may confound the results of the study, interfere with the patient's participation, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From randomization to time of first progression or death from any cause, whichever came first, assessed up to 5 years

SECONDARY OUTCOMES:
Overall survival (OS) | From randomization to the date of death from any cause, assessed up to 5 years
cancer-specific survival | From randomization to the date of death due to ovarian cancer, assessed up to 5 years
Treatment-related adverse events | From randomization up to the end of treatment plus 6 weeks
  assessed by CTCAE ver.5.0
Health-related quality of life (QLQ C30) | Over the 5 year surveillance period
  assessed by EEuropean Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Score 30 (QLQ-C30)
Health-related quality of life (QLQ OV28) | Over the 5 year surveillance period
  assessed by European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Ovarian Cancer Module (QLQ-OV28)
Health-related quality of life (EQ-5D-5L) | Over the 5 year surveillance period
  assessed by the 5-level EQ-5D version (EQ-5D-5L)
Cost-effectiveness analysis | At time of completion of 5-year surveillance period
  assessed by Quality-Adjusted Live Years (QALYs)

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Myong Cheol Lim, Goyang-si, Gyeonggi-do
  - Ewha Womans University Mokdong Hospital, Seoul
  - Korea University Anam hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim JH, Park E, Park SY, Lim MC. A randomized, multicenter, open-label phase III trial of cytoreductive surgery and hyperthermic intraperitoneal chemotherapy in platinum-resistant recurrent ovarian cancer: a rationale and study design of the KOV-HIPEC-02 trial. Int J Gynecol Cancer. 2025 Apr;35(4):101630. doi: 10.1016/j.ijgc.2025.101630. Epub 2025 Jan 9. PMID 39955184